CLINICAL TRIAL: NCT06413095
Title: Pembrolizumab Alone and in Combination(s) With MK-0482 and MK-4830 Via Intratumoral Injection in Patients With Head and Neck Squamous Cell Carcinoma or Soft Tissue Sarcoma Prior to Planned Surgical Intervention
Brief Title: PBI-MST-01 (NCT04541108) Substudy MSD-03: Intratumoral Microdosing of Pembrolizumab Alone and With MK-0482 or MK-4830 in HNSCC or STS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MST01-MSD-03; PBI-MST-01 (Other: Presage Biosciences)
Record Dates: First submitted 2024-04-01; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Soft Tissue Sarcoma
Keywords: HNSCC; head and neck cancer; head and neck squamous cell carcinoma; STS; soft tissue sarcoma; intratumoral microdosing; microdose injection; microdosing; in vivo oncology; tumor microenvironment; multiplexed immunohistochemistry; pharmacodynamic biomarkers; CIVO; master protocol; precision oncology; spatial biology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Sarcoma; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an exploratory clinical trial to evaluate intratumoral mechanistic effects of novel and approved agents on intact human tumors. This is a cohort substudy of a Master Protocol (PBI-MST-01, NCT04541108) framework, under which comparisons will not be made between substudy cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Alone or in Combination with MK-0482 or MK-4830 (Experimental): Patient with HNSCC or STS with surface accessible lesions who are scheduled for tumor or regional node dissection as part of their standard treatment will be injected two to four days prior to surgery using the CIVO device. Each needle of the CIVO device will deliver up to 8.3 microliters of solution, including a vehicle control (sterile saline) or subtherapeutic microdoses of pembrolizumab as a single agent or in combination with MK-0482 or MK-4830. Each microdose is simultaneously injected in a columnar fashion through each of 5 or 8 needles by the CIVO Micodose Injection Device (MID) into a single solid tumor or effaced metastatic lymph node.
  Interventions: Biological: Pembrolizumab; Combination Product: MK-0482 + Pembrolizumab; Combination Product: MK-4830 + Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Intratumoral microdose injection by the CIVO device.
  Other Names: Keytruda, MK-3475
Combination Product: MK-0482 + Pembrolizumab — Intratumoral microdose injection by the CIVO device.
Combination Product: MK-4830 + Pembrolizumab — Intratumoral microdose injection by the CIVO device.

SUMMARY:
This is a multi-center, open-label, Phase 0 substudy designed to evaluate the ability of pembrolizumab, alone and in combination with MK-0482 or MK-4830, to elicit pharmacodynamic changes suggestive of antitumor immune activation within the native tumor microenvironment (TME) following intratumoral microdosing via the CIVO device in patients with surface accessible Head and Neck Squamous Cell Carcinoma (HNSCC) or Soft Tissue Sarcoma (STS) lesion(s) who are scheduled for tumor and/or regional node dissection as part of their standard treatment.

DETAILED DESCRIPTION:
The CIVO Microdose Injection Device (MID) simultaneously delivers multiple drugs and drug combinations (up to 8), each in microdose amounts, into a single patient tumor and enables comparisons of the resulting biomarker responses that occurred while that tumor was still in the native microenvironment. The microdose injection procedure is conducted ahead of the patient's scheduled surgical intervention and localized biomarker responses are then evaluated in the injected tumor tissue following surgery. This enables assessments of drug-induced changes to the tumor, stroma, and local immune cells within the unique landscape of each individual patient and their respective tumor genomic profile and immune system functional status. CIVO is a research tool used only to assess the responses of tumor cells and other cell populations with the TME following intratumoral administration of drug microdoses; it is not a therapeutic device.

MK-0482, MK-4830, and pembrolizumab have distinct mechanisms of action (MOAs) that affect the TME, including relief of immune suppression and enhanced T-cell activation. Surgery is the standard primary treatment for most patients with STS, and surgical intervention of the primary tumor and cervical lymph node dissection may be recommended for patients with HNSCC. Dysfunction of the immune system (e.g., immune evasion, expression of suppressive immune checkpoint receptors, etc.) plays a major role in the development and progression of HNSCC and STS. Therefore, in this Phase 0 study, the ability of pembrolizumab, alone and in combination with MK-0482 or MK-4830, to elicit pharmacodynamic changes suggestive of antitumor immune activation within the native TME in patients with HNSCC or STS will be assessed. Pembrolizumab, alone and in combination with MK-0482 or MK-4830, will be injected in microdose quantities at tumor sites in HNSCC or STS patients with a surface accessible lesion who are scheduled for tumor and/or regional node dissection as part of their standard treatment. Injected tumors will be resected as per surgical standard of care following 2 to 4 days in situ exposure. Thereafter, the CIVO-injected portion of the tissue will be analyzed for localized response at sites of drug exposure in the TME.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of HNSCC or STS.
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary tumor, recurrent tumor, or metastatic lymph node) of at least approximately 2.5 cm in the shortest diameter that is surface accessible for CIVO injection that contains viable minimum tissue volume and characteristics (e.g., based on clinical evaluation, available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports indication lesion with appropriate viable tumor volume, without excessive cysts or necrosis) and for which there is a planned surgical intervention.
6. Female patients who:

   * Are postmenopausal for at least one year before the screening visit, OR
   * Are surgically sterile, OR
   * Are of childbearing potential who agree to practice a highly effective method of contraception from the time of signing the Informed Consent Form (ICF) through up to 120 days after the tumor injection procedure OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating ova during study participation.

   Male patients, even if surgically sterile (i.e., status post-vasectomy), who:
   * Agree to practice effective barrier contraception from the time of signing the ICF and during study participation OR agree to completely abstain from heterosexual intercourse.
   * Agree to refrain from donating sperm during study participation.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

1. Patients who have received neoadjuvant therapy associated with the surgical intervention described in Inclusion Criterion #5 within 6 months of the CIVO injection procedure.
2. Tumors near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
3. Female patients who are:

   * Both lactating and breastfeeding, OR
   * Have a positive beta human chorionic gonadotropin (beta-hCG) pregnancy test at screening verified by the Investigator.
4. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
5. Patients with a history of concurrent second cancers requiring active, ongoing systemic treatment. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
6. Patients with a diagnosis of immunodeficiency.
7. Patients with known HIV/AIDS with uncontrolled viral load and CD4 less than 200, or those with concurrent active hepatitis B (defined as HBsAg positive or detectable HBV DNA) or hepatitis C (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Note: HIV infected participants with a history of Kaposi's sarcoma or Multicentric Castleman's Disease are excluded. Hepatitis B and C screening tests are not required unless:

   * Patient has a known history of hepatitis B/C infection
   * Mandated by local health authority
8. Patients that have received a live or live-attenuated vaccine within 4 weeks of the baseline/screening visit.
9. Use of any of the following ≤ 2 weeks prior to CIVO injection:

   1. Chronic systemic immunosuppressive therapy or corticosteroids (in dosing exceeding 10 mg daily of prednisone equivalent). Intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular injection), or steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication) are exceptions to this criterion.
   2. Biological response modifiers for treatment of active autoimmune disease.
   3. Hematopoietic growth factors.
10. Patients who have received prior treatment with radiation or systemic therapy (e.g., cytotoxic chemotherapy, targeted agents, or checkpoint inhibitor immunotherapy, etc.), or have participated in a study of an investigational device within 6 months of the CIVO injection procedure. Note: Participants must have recovered from all radiation-related toxicities, must not require corticosteroids, and must not have had radiation pneumonitis.
11. Patients who have a history of (noninfectious) pneumonitis that required steroids or have current pneumonitis.
12. Patients who have had allogenic tissue/solid organ transplant.
13. Patients who have had severe hypersensitivity (≥Grade 3) to pembrolizumab, MK-4830, MK-0482, or any of their excipients.
14. Patients with an active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Quantification of Immune Cell Biomarkers by Immunohistochemistry (IHC), In Situ Hybridization (ISH), and/or Spatial Biology Platforms | 2 to 4 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumor microenvironment around injection sites in resected patient samples by IHC, ISH, or spatial biology platforms. An aggregate analysis of this quantification may be done across patient samples in each substudy to evaluate trends in tumor response. The biomarkers evaluated may include, but are not limited to, markers associated with macrophage polarization states (e.g., CD163), markers of infiltrating T cells (e.g., CD8/Granzyme B), and proinflammatory cytokines (e.g., interferon gamma).

SECONDARY OUTCOMES:
Incidence of reported Adverse Events and/or Adverse Device Effects [Safety and Tolerability] | Up to 28 days after microdose injection
  Safety of the microdose injection procedure and injected content will be assessed by quantification of the frequency, intensity, and relatedness of all reported Adverse Events and/or Adverse Device Effects.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Presage Biosciences
Locations (11):
- United States (11):
  - UC Davis, Sacramento, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - LSU Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - UC Health, Cincinnati, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Medical Center, Charleston, South Carolina
  - UT Health Houston, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derry JMJ, Burns C, Frazier JP, Beirne E, Grenley M, DuFort CC, Killingbeck E, Leon M, Williams C, Gregory M, Houlton J, Clayburgh D, Swiecicki P, Huszar D, Berger A, Klinghoffer RA. Trackable Intratumor Microdosing and Spatial Profiling Provide Early Insights into Activity of Investigational Agents in the Intact Tumor Microenvironment. Clin Cancer Res. 2023 Sep 15;29(18):3813-3825. doi: 10.1158/1078-0432.CCR-23-0827. PMID 37389981
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571